CLINICAL TRIAL: NCT00827827
Title: Strength Training for Skeletal Muscle Adaptation After Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B6737-R; H30631 (Other: Baltimore VAMC)
Record Dates: First submitted 2009-01-22; First posted 2009-01-23 (Estimated); Results first posted 2015-01-19 (Estimated); Last update posted 2018-07-09 (Actual); Status verified 2018-06

CONDITIONS: Stroke
Keywords: Stroke; Exercise; Strength Training; Skeletal Muscle; Insulin Sensitivity
MeSH Terms: conditions — Stroke; Motor Activity; Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm 1 (Experimental): Participants in this group undergo lower-extremity strength training on three pneumatic resistance machines (Keiser Leg Press, Keiser Leg Extension, and Keiser Leg Curl). Training sessions happen 3 times per week (M,W,F) and last approximately 45 minutes to 1 hour. Participants in this group exercise each limb individually to account for the large discrepancies in strength between legs in stroke survivors.
  Interventions: Other: Exercise- Strength Training
- Arm 2 (Active Comparator): Participants in this group receive equal exposure to study staff compared with the experimental ST group (approximately 45 minutes to 1 hour 3 times per week). Exercise sessions for this group involve a full battery of active and passive...upper and lower body...stretching and range of motion exercises performed on raised padded tables.
  Interventions: Other: Exercise- Stretching Control

INTERVENTIONS:
Other: Exercise- Strength Training — 3x per week lower-extremity ST lasting approximately 45 minutes to 1 hour.
  Arms: Arm 1
Other: Exercise- Stretching Control — 3x per week upper and lower body stretching mixed with active and passive range of motion exercises
  Arms: Arm 2

SUMMARY:
Chronically disabled stroke survivors experience accelerated skeletal muscle atrophy and other detrimental changes to muscle and surrounding tissues on the paretic side. This unilateral tissue-level damage contributes to worsening disability and insulin resistance. This VA Merit Award will advance the investigators' understanding of the potential for strength training (ST) to reverse stroke-related muscle abnormalities to improve metabolic health, strength, and function. It will be the first study to thoroughly investigate the effects of ST on muscle atrophy, intramuscular fat, muscle fiber characteristics, capillary density and insulin sensitivity after stroke.

DETAILED DESCRIPTION:
This study investigates the hypothesis that a novel, high intensity, high repetition ST program will improve abnormalities in paretic and non-paretic leg muscle volume and composition compared to an attention-matched control regimen of supervised stretching over a 3-month intervention period in those disabled by stroke. The investigators further hypothesize that ST-induced skeletal muscle adaptation will translate into improved insulin sensitivity, strength, and function in this population. The specific objectives are to: 1) Determine the effects ST compared to a control intervention on paretic and non-paretic abnormalities in skeletal muscle volume, intramuscular fat, muscle fiber distribution, muscle capillary density, and muscle inflammation in chronically disabled stroke survivors. 2) Determine the effects ST compared to a control intervention on insulin sensitivity in stroke survivors, and whether structural and cellular skeletal muscle mechanisms contribute to improvements in insulin sensitivity after ST. 3) Determine the effects ST compared to a control intervention on physical function (strength, walking speed and balance) in stroke survivors, and whether structural skeletal muscle mechanisms predict ST-induced functional improvement.

The project design consists of 4 phases over 5 months for stroke participants enrolled in either of the two intervention arms (ST vs. CONTROL). During phase 1 the investigators will screen and consent chronic stroke patients with residual gait deficits. Phase 2 (3 weeks) will consist of baseline testing that includes dual energy X-ray absorptiometry (DEXA) scanning, bilateral CT scanning of the legs, bilateral vastus lateralis muscle biopsies, strength testing, timed walks, balance measurements, oral glucose tolerance testing, and hyperglycemic clamp testing. Following completion of baseline testing, volunteers are to be randomized to ST or the CONTROL group. Phase 3 (Intervention Phase, 3 months) will begin with 2 sessions of acclimatization for those assigned to the ST group. ST will then be progressed to 2 sets of 20 repetitions on each leg on each machine (Keiser Leg Press, Leg Extension, Leg Curl) with gradual increases in resistance over 3 months. Those in the CONTROL group will receive equal exposure to health care personnel in the Baltimore VA Exercise facility, performing a full battery of upper and lower body passive and active stretching exercises at each intervention session. In Phase 4 all baseline testing and laboratory analyses will be repeated.

Developing evidence-based therapies to combat skeletal muscle deterioration is highly relevant for chronically disabled stoke survivors. There is mounting evidence that current models of post-stroke rehabilitation are not optimal for maximizing recovery of muscle mass, strength, and metabolic health. The proposed research will develop new insight into the utility of progressive ST for reversing detrimental changes to gross muscle composition, muscle molecular phenotype, muscle inflammation, and muscle capillarization. Changes to any or all of these muscle parameters should have measurable impact on both whole body insulin sensitivity and function. Collectively, the results from this trial may change the current standard of care for stroke survivors by providing evidenced reasons for augmenting physical therapists' treatments, allowing more intense and diverse therapy sessions for maintenance of skeletal muscle.

ELIGIBILITY:
Inclusion Criteria:

* Stroke greater than 6 months prior with residual hemiparetic gait in women or men aged 40-85 years
* Completion of all regular post-stroke physical therapy
* Adequate language and neurocognitive function to participate in testing and training and to give adequate informed consent

Exclusion Criteria:

* Alcohol consumption greater than 3 oz. liquor, or 3 x 4 oz glasses of wine, or 3 x 12 oz. beers per day, by self-report
* clinical history of:

  * unstable angina
  * recent (less than 3 months) myocardial infarction or congestive heart failure (NYHA category II)
  * hemodynamically significant valvular dysfunction
  * peripheral arterial occlusive disease (PAOD) with claudication
  * major orthopedic, chronic pain, or non-stroke neuromuscular disorders restricting exercise
  * pulmonary or renal failure
  * poorly controlled hypertension (greater than 190/110)
  * recent hospitalization for severe disease or surgery
  * severe or global receptive aphasia which confounds reliable testing and training
* Allergy to lidocaine
* Known muscle disorder
* Taking Coumadin or Lovenox (contraindication for muscle biopsies)
* Dementia
* Untreated major depression

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2009-04-01 (Actual); Primary Completion 2013-08-31 (Actual); Study Completion 2018-06-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frederick M Ivey, PhD, Principal Investigator — Baltimore VA Medical Center VA Maryland Health Care System, Baltimore, MD
Locations (1):
- Baltimore VA Medical Center VA Maryland Health Care System, Baltimore, MD, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ivey FM, Prior SJ, Hafer-Macko CE, Katzel LI, Macko RF, Ryan AS. Strength Training for Skeletal Muscle Endurance after Stroke. J Stroke Cerebrovasc Dis. 2017 Apr;26(4):787-794. doi: 10.1016/j.jstrokecerebrovasdis.2016.10.018. Epub 2016 Nov 16. PMID 27865696
- [Result] Ivey FM, Ryan AS. Resistive training improves insulin sensitivity after stroke. J Stroke Cerebrovasc Dis. 2014 Feb;23(2):225-9. doi: 10.1016/j.jstrokecerebrovasdis.2012.12.014. Epub 2013 Jan 22. PMID 23352685

RESULTS

PARTICIPANT FLOW:
Groups:
- Strength Training: Participants in this group undergo lower-extremity strength training on three pneumatic resistance machines (Keiser Leg Press, Keiser Leg Extension, and Keiser Leg Curl). Training sessions happen 3 times per week (M,W,F) and last approximately 45 minutes to 1 hour. Participants in this group exercise each limb individually to account for the large discrepancies in strength between legs in stroke survivors.
  Exercise- Strength Training: 3x per week lower-extremity ST lasting approximately 45 minutes to 1 hour.
- Stretching Control: Participants in this group receive equal exposure to study staff compared with the experimental ST group (approximately 45 minutes to 1 hour 3 times per week). Exercise sessions for this group involve a full battery of active and passive...upper and lower body...stretching and range of motion exercises performed on raised padded tables.
  Exercise- Stretching Control: 3x per week upper and lower body stretching mixed with active and passive range of motion exercises
Period: Overall Study
Arm/Group | Strength Training | Stretching Control
Started | 22 | 16
Completed | 14 | 16
Not Completed | 8 | 0
Not completed — Lost to Follow-up | 3 | 0
Not completed — Fall at home- hospitalization | 1 | 0
Not completed — Another cerebrovascular accident (CVA) | 1 | 0
Not completed — Gout | 1 | 0
Not completed — Transportation issues | 1 | 0
Not completed — Burned with water at home | 1 | 0

BASELINE CHARACTERISTICS:
Population: Disabled stroke survivors
Groups:
- Total: Total of all reporting groups
Arm/Group | Strength Training | Stretching Control | Total
Number analyzed (Participants) | 22 | 16 | 38
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 19 | 14 | 33
  >=65 years | 3 | 2 | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.9 (11.5) | 55.2 (8.7) | 56.2 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 4 | 10
  Male | 16 | 12 | 28
Region of Enrollment [Number; unit: participants]
  United States | 22 | 16 | 38

OUTCOME MEASURES:

1. Primary Outcome: Change in 1-repetition Maximum (RM) Muscle Strength (Leg Press, Paretic Side)
Time Frame: Baseline, 3 months
Population: All participants for whom strength measurements were recorded at Baseline and 3 months
Measure: Mean (Standard Error); unit: lbs
Arm/Group | Strength Training | Stretching Control
Number analyzed (Participants) | 14 | 16
lbs | 126.1 (22.2) | 11.3 (14.6)

2. Primary Outcome: Change in 1-RM Muscle Strength (Leg Press, Non-Paretic Side)
Time Frame: Baseline, 3 months
Population: All participants for whom strength measurements were recorded at Baseline and 3 months
Measure: Mean (Standard Error); unit: lbs
Arm/Group | Strength Training | Stretching Control
Number analyzed (Participants) | 14 | 16
lbs | 93.2 (26.1) | 22.7 (16.4)

3. Primary Outcome: Change in 1-RM Muscle Strength (Leg Extension, Paretic Side)
Time Frame: Baseline, 3 Months
Population: All participants for whom strength measurements were recorded at Baseline and 3 months
Measure: Mean (Standard Error); unit: lbs
Arm/Group | Strength Training | Stretching Control
Number analyzed (Participants) | 14 | 16
lbs | 28.6 (4.3) | 3.4 (2.4)

4. Primary Outcome: Change in 1-RM Muscle Strength (Leg Extension, Non-Paretic Side)
Time Frame: Baseline, 3 Months
Population: All participants for whom strength measurements were recorded at Baseline and 3 months
Measure: Mean (Standard Error); unit: lbs
Arm/Group | Strength Training | Stretching Control
Number analyzed (Participants) | 13 | 16
lbs | 20.8 (0.4) | 0.4 (2.6)

5. Primary Outcome: Change in Leg Muscle Endurance (Paretic Side)
Description: Tests how training impacts the total number of submaximal repetitions a participant can perform according to standardized cadence (at the same absolute level of resistance, pre and post).
Time Frame: Baseline, 3 Months
Population: All participants for whom muscle endurance measurements were recorded at Baseline and 3 months
Measure: Mean (Standard Error); unit: repetitions
Arm/Group | Strength Training | Stretching Control
Number analyzed (Participants) | 14 | 15
repetitions | 27.4 (4.5) | 2.0 (2.1)

6. Primary Outcome: Change in Leg Muscle Endurance (Non-Paretic Side)
Description: as for outcome 5
Time Frame: Baseline, 3 months
Population: All participants for whom muscle endurance measurements were recorded at Baseline and 3 months
Measure: Mean (Standard Error); unit: repetitions
Arm/Group | Strength Training | Stretching Control
Number analyzed (Participants) | 14 | 15
repetitions | 27.5 (5.0) | 1.8 (1.8)

7. Primary Outcome: Change in 6-minute Walk Distance
Time Frame: Baseline, 3 Months
Population: All participants for whom 6-minute walk distance was recorded at Baseline and 3 months
Measure: Mean (Standard Error); unit: feet
Groups:
- Stretching Controls: Participants in this group receive equal exposure to study staff compared with the experimental ST group (approximately 45 minutes to 1 hour 3 times per week). Exercise sessions for this group involve a full battery of active and passive...upper and lower body...stretching and range of motion exercises performed on raised padded tables.
  Exercise- Stretching Control: 3x per week upper and lower body stretching mixed with active and passive range of motion exercises
Arm/Group | Strength Training | Stretching Controls
Number analyzed (Participants) | 13 | 16
feet | 132.3 (48.3) | -2.1 (21.6)

8. Primary Outcome: Change in 10 Meter Walking Speed (Self-Selected)
Time Frame: Baseline, 3 months
Population: All participants for whom 10 Meter walking Speed (Self-Selected) was recorded at Baseline and 3 months
Measure: Mean (Standard Error); unit: meters/ second
Arm/Group | Strength Training | Stretching Controls
Number analyzed (Participants) | 14 | 16
meters/ second | 0.16 (0.09) | 0.03 (0.06)

9. Primary Outcome: Change in 10 Meter Walking Speed (Fastest)
Time Frame: Baseline, 3 Months
Population: All participants for whom 10 Meter walking Speed (Fastest-Safe) was recorded at Baseline and 3 months
Measure: Mean (Standard Error); unit: meters/ second
Arm/Group | Strength Training | Stretching Controls
Number analyzed (Participants) | 13 | 14
meters/ second | 0.24 (0.10) | 0.09 (0.08)

10. Primary Outcome: Change in Peak Aerobic Capacity (VO2 Peak)
Time Frame: Baseline, 3 Months
Population: All participants for whom Peak Aerobic Capacity was recorded during Graded Treadmill Test at Baseline and 3 months
Measure: Mean (Standard Error); unit: mls/kg/min
Arm/Group | Strength Training | Stretching Controls
Number analyzed (Participants) | 14 | 15
mls/kg/min | 1.2 (0.6) | -0.4 (0.5)

11. Primary Outcome: Change in Berg Balance Scale
Description: This measure is a 14 item scale, with each item scored (0-4) and summed for a maximum score of 56 points. Range is 0-56 and higher values represent a better outcome.
Time Frame: Baseline, 3 months
Population: All participants for whom a Berg Score was recorded at Baseline and 3 months
Measure: Mean (Standard Error); unit: Scores on a scale
Arm/Group | Strength Training | Stretching Control
Number analyzed (Participants) | 14 | 16
Scores on a scale | 0.3 (0.6) | -0.1 (0.5)

12. Primary Outcome: Change in Paretic Limb Step Time (Self-Selected)
Description: This and other measures come from Instrumented Walkway (Gait Rite)
Time Frame: Baseline, 3 months
Population: All participants for whom measurement was recorded at Baseline and 3 months
Measure: Mean (Standard Error); unit: seconds
Arm/Group | Strength Training | Stretching Control
Number analyzed (Participants) | 13 | 11
seconds | -0.04 (0.03) | -0.03 (0.03)

13. Primary Outcome: Change in Paretic Limb Step Time (Fastest)
Description: This and other measures come from Instrumented Walkway (Gait Rite)
Time Frame: Baseline, 3 Months
Population: All participants for whom measurement was recorded at Baseline and 3 months
Measure: Mean (Standard Error); unit: seconds
Arm/Group | Strength Training | Stretching Control
Number analyzed (Participants) | 13 | 10
seconds | 0.00 (0.03) | 0.00 (0.02)

14. Primary Outcome: Change in Non-Paretic Limb Step Time (Self-Selected)
Description: This and other measures come from Instrumented Walkway (Gait Rite)
Time Frame: Baseline, 3 months
Population: All participants for whom measurement was recorded at Baseline and 3 months
Measure: Mean (Standard Error); unit: seconds
Arm/Group | Strength Training | Stretching Control
Number analyzed (Participants) | 13 | 11
seconds | -0.01 (0.02) | -0.07 (0.05)

15. Primary Outcome: Change in Non-Paretic Limb Step Time (Fastest)
Description: This and other measures come from Instrumented Walkway (Gait Rite)
Time Frame: Baseline, 3 Months
Population: All participants for whom measurement was recorded at Baseline and 3 months
Measure: Mean (Standard Error); unit: seconds
Arm/Group | Strength Training | Stretching Control
Number analyzed (Participants) | 13 | 10
seconds | -0.01 (0.02) | -0.01 (0.01)

16. Primary Outcome: Change in Paretic Limb Step Length (Self-Selected)
Description: This and other measures come from Instrumented Walkway (Gait Rite)
Time Frame: Baseline, 3 Months
Population: All participants for whom measurement was recorded at Baseline and 3 months
Measure: Mean (Standard Error); unit: cm
Arm/Group | Strength Training | Stretching Control
Number analyzed (Participants) | 13 | 11
cm | 4.0 (1.5) | 1.1 (2.8)

17. Primary Outcome: Change in Paretic Limb Step Length (Fastest)
Description: This and other measures come from Instrumented Walkway (Gait Rite)
Time Frame: Baseline, 3 months
Population: All participants for whom measurement was recorded at Baseline and 3 months
Measure: Mean (Standard Error); unit: cm
Arm/Group | Strength Training | Stretching Control
Number analyzed (Participants) | 13 | 10
cm | 3.8 (2.1) | 0.9 (2.7)

18. Primary Outcome: Change in Non-Paretic Limb Step Length (Self-Selected)
Description: This and other measures come from Instrumented Walkway (Gait Rite)
Time Frame: Baseline, 3 Months
Population: All participants for whom measurement was recorded at Baseline and 3 months
Measure: Mean (Standard Error); unit: cm
Arm/Group | Strength Training | Stretching Control
Number analyzed (Participants) | 13 | 11
cm | 3.8 (1.4) | 0.3 (2.1)

19. Primary Outcome: Change in Non-Paretic Limb Step Length (Fastest)
Description: This and other measures come from Instrumented Walkway (Gait Rite)
Time Frame: Baseline, 3 Months
Population: All participants for whom measurement was recorded at Baseline and 3 months
Measure: Mean (Standard Error); unit: cm
Arm/Group | Strength Training | Stretching Control
Number analyzed (Participants) | 13 | 10
cm | 4.6 (1.9) | -0.4 (3.0)

ADVERSE EVENTS:
Arm/Group | Strength Training | Stretching Control
Serious Adverse Events (participants affected / at risk) | 2/22 | 2/16
Other Adverse Events (participants affected / at risk) | 3/22 | 9/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Strength Training (N=22) | Stretching Control (N=16)
fell at home (General disorders) | 1 (1) | 1 (1) — required hospitalization.
hypotensive episode (General disorders) | 1 (1) | 0 (0) — following a training session. Further evaluation indicated the need for hospital admission.
choked on a pill at home (General disorders) | 0 (0) | 1 (1) — went to the ER where he was held overnight
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Strength Training (N=22) | Stretching Control (N=16)
hypotensive event (General disorders) | 1 (1) | 2 (2) — not requiring hospitalization
falls outside of training/ testing sessions (General disorders) | 0 (0) | 5 (5) — none requiring hospitalization
muscle strain (General disorders) | 1 (1) | 1 (1) — not requiring hospitalization
gout flare-up (General disorders) | 0 (0) | 1 (1) — no hospitalization but treated by PCP
adverse reaction to lidocaine during muscle biopsy (General disorders) | 1 (1) | 0 (0) — symptoms resolved after 40 minutes

LIMITATIONS AND CAVEATS:
Scanning results and muscle biopsy outcomes are still pending and won't be available for some time.

Numbers of participants qualifying for and agreeing to metabolic testing will be too low to yield reportable results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes